CLINICAL TRIAL: NCT05551858
Title: A Phase 1/2 Trial to Test the Safety of a CCK Receptor Antagonist, Proglumide, in Management of Chronic Pancreatitis Symptoms and Pain for 12 to 24 Months
Brief Title: Role of a CCK Receptor Antagonist Proglumide in Management of Chronic Pancreatitis
Acronym: ProCP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5063
Record Dates: First submitted 2022-09-01; First posted 2022-09-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Safety Issues; Pain; Pancreas Fibrosis
Keywords: Cholecystokinin; Pain; Proglumide; Diabetes; Pancreatitis
MeSH Terms: conditions — Pain; Diabetes Mellitus; Pancreatitis | interventions — Proglumide

STUDY DESIGN:
Intervention Model Description: Part-1 Single group Part-2 crossover
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part-2 First 12- weeks includes 1:1 drug versus placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Arm 1. Placebo for first 12 weeks. Placebo is a fiber filler called Avicel and is given by mouth three times daily.
  Note: After 12 weeks on placebo, these subjects will receive proglumide 400 mg orally three times daily open labeled for 12 additional weeks.
  Interventions: Drug: Placebo
- Proglumide (Experimental): Proglumide therapy 400 mg by mouth three times daily for 12 weeks in a blinded fashion followed by continued proglumide 400 mg by mouth three times daily for 12 additional weeks in an open labeled fashion. Hence this arm receives proglumide for a total of 24 weeks.
  Interventions: Drug: Proglumide

INTERVENTIONS:
Drug: Proglumide — (CAS: 6620-60-6.)
  Other Names: Milid
  Arms: Proglumide
Drug: Placebo — Avicel fiber filled capsule taken by mouth three times daily
  Arms: Placebo

SUMMARY:
Chronic pancreatitis is a rare but debilitating condition associated with chronic abdominal pain, diarrhea, diabetes, and an 8-fold increased risk for the development of pancreatic cancer. Unfortunately, there is no available treatment to prevent the progression of chronic pancreatitis, and most subjects require narcotic medications to control the pain. A receptor protein call the CCK-B receptor becomes activated in chronic pancreatitis and is in part responsible for the scar tissue or fibrosis that occurs and responsible for the cancer risk. In mice with chronic pancreatitis, the inflammation and damage was reversed with an old drug called proglumide that blocks the activation of the CCK-B receptor. Proglumide has also been shown to possibly reduce pain.

This protocol involved a 2-Part study to test the safety of oral proglumide in those with confirmed chronic pancreatitis and the second goal is to determine if proglumide improves pain and function of the pancreas. Part-1 is an open-labelled Lead-in Study of N=8 subjects over a 12-week treatment period. Part-2 is a randomized double blind pseudo cross over study where subjects will be treated in Arm A (placebo for 12 weeks followed by 12 weeks of proglumide) and Arm B ( proglumide for 24 weeks).

DETAILED DESCRIPTION:
Part-1 open labeled:

At screening, laboratory tests will be performed including: Liver profile, Basic chemistry with renal profile, CBC & platelets, serum lipase levels, HgbA1C, and CRP. A history and physical exam, and the numeric Pain scale diary will be provided. Subjects will be asked to record their worse pain score on a scale of 0 to 10 for each 24 hours over a seven day period. An average pain score of 5 is required for eligibility. Those meeting enrolment criteria according to lab and clinical criteria will go into the next phase.

Observation phase: Within 14 days ± 3 days, subjects that meet the inclusion criteria will have baseline Pain surveys done (Patient-Reported Outcomes Measurement Information Systems- PROMIS and COMPAT-SF) and keep a diary using the numeric pain scale (NPS) daily to record their maximum pain score for each day. The observation period will be 4 weeks. After completing the observation phase, subjects will come to CRU for the baseline visit. The pain surveys can be given to the subjects at the screening visit or sent to the subjects and completed at their home or with the assistance of the Study Coordinator on the Phone.

Baseline: At the baseline visit in the CRU, Pain diaries will be collected from the observation phase and repeat Pain Surveys will be performed (see outcomes below) and Basic chemistry with renal profile, CBC & platelets, serum lipase levels, HgbA1C, and CRP will be drawn. A history and physical exam will be performed and one red-top blood tube collected and serum frozen for a biomarker and cytokine panels. A 32-day supply of proglumide (#96) will be dispensed with instructions to administer 400mg po TID. A diary for recording pain, medication diary, recording proglumide consumption and any adverse effects will be dispensed and a follow-up appointment scheduled in 4 weeks ± 4 days.

Follow-up visits: (4 week intervals ± 3 days) Subjects will return at weeks 4, 8, 12 and 16 and bring their daily NPS diaries and medication records and bottles for review and accountability. Pain Surveys will be completed at the visits with the assistance of the study coordinator. Concomitant medications and adverse events will be reviewed. Repeat laboratory tests (same as screening) will be repeated. At weeks 4 and 8 another month's supply of proglumide will be dispensed and new diaries. At week-12 a repeat research blood tube will be collected for the biomarker investigation and for proglumide blood level analysis if needed. At weeks 12 and 16 no medication will be dispensed. The week-16 is the follow-up safety visit off medication. At each follow-up visit, subjects should also be evaluated for signs and symptoms of gallbladder pathology.

Part-2 Randomized placebo controlled pseudo crossover:

The second Part will be a randomized placebo-controlled pseudo-crossover study with N=12 subjects in each arm. Part 2 will not start until all subjects complete Part 1 and there are no safety issues. Note: Subjects that participated in Part 1 may be eligible to participate in Part 2 if the subjects meet all the inclusion criteria. A 90-day washout is required off proglumide.

Screening: Screening for the Part 2 study will be the same as that for Part 1 above. There will be no observation untreated phase in this Part.

Baseline visit: Within 14±3 days after subjects are consented, screened and meet the inclusion criteria, the subject will come to the Clinical research Unit (CRU) at 1 PHC for the baseline visit. Subjects will undergo MRI imaging at this visit or after the subject meets the inclusion criteria within the 14 days. If an abdominal MRI was done within the past 3 months with contrast and imaging of the pancreas, a repeat MRI will not be repeated. At the baseline visit the investigational pharmacist will perform the blinded randomization and either a 45-day supply of proglumide (#135) will be dispensed with instructions to administer 400mg po TID or a 45-day supply of placebo to take po TID. Pain Surveys will be performed (see outcomes below) and basic chemistry with renal profile, CBC & platelets, serum lipase levels, HgbA1C, and CRP will be drawn. A history and physical exam will be performed and one red-top blood tube collected and serum frozen for a biomarker and cytokine panels. A diary for recording pain, medication diary, recording proglumide consumption and any adverse effects will be dispensed and a follow-up appointment scheduled in 6 weeks ± 4 days.

Follow-up visits: (every 6 weeks ± 3 days); follow up visits will occur at weeks 6, 12, 18, and 24. Pain Surveys will be completed at the visits with the assistance of the study coordinator. Concomitant medications and adverse events will be reviewed. Drug accountability will be done. Repeat laboratory tests will be done: Liver profile, Basic chemistry with renal profile, CBC & platelets, serum lipase levels, HgbA1C, and CRP. AT week 6 the pharmacy will dispense either proglumide or placebo according to the subject's randomization. Leftover capsules may be redispensed to the subject. AT week-12, all medication will be returned to the pharmacy and a new Rx will be dispensed to all subjects containing active drug, proglumide 400 mg to take po TID. At week-12 another research biomarker / proglumide blood tube will be collected and an MRI (preferably at the same location as Baseline) will be done to evaluate the pancreas. At week 18, another research tube will be collected for research biomarker panel/ proglumide blood analysis and all medication will be returned.

Safety termination visit: Four weeks after completing the treatment phase subjects will return for a safety check. Symptoms will be reviewed; the Numeric pain score assessed; and Laboratory tests will be drawn (Liver profile, Basic chemistry with renal profile, CBC & platelets, serum lipase levels, HgbA1C, and CRP).

ELIGIBILITY:
Subjects are eligible with a history of chronic pancreatitis as defined by the Cambridge radiographic classification with abnormal pancreatic side branches but without main pancreatic duct obstructing calcifications.

Inclusion Criteria:

* Males or females age 18 to 75 years of age
* Clinical symptoms of chronic pancreatitis
* Plus confirmation of chronic pancreatitis with imaging (Cambridge classification), EUS, biopsy, or fecal elastase <200µg/g, or abnormal 72 hr fecal fat and radiographic evidence of CP.
* Pain not adequately controlled with medications
* Pain of at least 5 on a numeric pain scale of 0-10
* Stable doses of anti-diabetic medication for at least 90 days prior to screening.
* Women of childbearing potential unless surgically sterile or using adequate contraception (either IUD, oral or deport contraceptive, or barrier plus spermicide).
* Both males and females must be willing and able to continue contraception to prevent pregnancy for 3 months after the completion of the study.

Exclusion Criteria:

* Currently abusing alcohol (more than three drinks in a day or more than seven drinks per week) or nonprescription drugs
* Pregnant or lactating, or unwilling to prevent pregnancy
* Renal insufficiency; CKD; GFR<60
* Unable to sign consent or maintain a diary
* Liver enzymes > 2x ULN, Hgb <8.5, Creat>2; HgbA1c>8
* Type 1 Diabetes
* Subjects with confirmed cirrhosis
* Evidence of active gallbladder disease or gallbladder dyskinesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood chemistry tests | 12 weeks of therapy
  Number of participants with abnormal chemistry blood tests at 12-weeks in placebo arm compared to treatment arm
Adverse events | 12 weeks of therapy
  Number of Adverse events according to the Common Toxicity criteria Version 5.0 occurring in proglumide-treated compared to placebo-treated groups

SECONDARY OUTCOMES:
Change in Pain Measurements from baseline to end of treatment with proglumide compared to Placebo | Baseline mean scores on a scale of 1 to 5 will be compared to scores at 12 weeks and 24 weeks
  Change in Pain score from baseline using the Patient-Reported Outcomes Measurement Information System (PROMIS Item Bank v1.1 - Pain Interference scale 1-5).
Change in Pain Measurements numeric score from baseline to end of treatment with proglumide compared to Placebo | Baseline mean scores compared to scores at 12 weeks and 24 weeks
  Change in mean pain scores on a scale of 0 to 10 at baseline to end of treatment using the Numeric Pain Scale (ranking of intensity of pain over 24 hr scored with a number from 0 or no pain to 10- severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Smith, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Funded by federal funds so required to share all information
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study complete and published
Access Criteria: Internet
URL: https://www.clinicaltrials.gov/

REFERENCES:
- [Result] Nadella S, Ciofoaia V, Cao H, Kallakury B, Tucker RD, Smith JP. Cholecystokinin Receptor Antagonist Therapy Decreases Inflammation and Fibrosis in Chronic Pancreatitis. Dig Dis Sci. 2020 May;65(5):1376-1384. doi: 10.1007/s10620-019-05863-5. Epub 2019 Oct 9. PMID 31598921